CLINICAL TRIAL: NCT06050460
Title: A Phase I Clinical Trial to Evaluate the Safety, Tolerance and Pharmacokinetics of A Broad-Spectrum Neutralizing Antibodies SA55 Injection of COVID-19 in Healthy Adults
Brief Title: SA55 Injection: a Potential Therapy for the Prevention and Treatment of COVID-19
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sinovac Life Sciences Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Sinovac Biotech Co., Ltd (Industry)
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: PRO-SA55-1001
Record Dates: First submitted 2023-08-26; First posted 2023-09-22 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The study will be blinded for all placebo controlled dose groups, ie, the principal investigator (PI), all clinical staff involved in the clinical study, the participants, and the study monitor will remain blinded, unless safety concerns or a regulatory requirement necessitate unblinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SA55 injection (Experimental): Cohort 1: 150mg; Cohort 2: 300mg; Cohort3: 600 mg; Cohort4: 900 mg
  Interventions: Drug: SA55 Injection
- Placebo for SA55 injection (Placebo Comparator): Cohort 1: 0mg; Cohort 2: 0mg; Cohort3: 0mg; Cohort4: 0mg
  Interventions: Other: Placebo for SA55 injection

INTERVENTIONS:
Drug: SA55 Injection — Novel coronavirus broad-spectrum neutralizing antibody SA55 injection
  Arms: SA55 injection
Other: Placebo for SA55 injection — Placebo for Novel coronavirus broad-spectrum neutralizing antibody SA55 injection
  Arms: Placebo for SA55 injection

SUMMARY:
In this first-in-humans dose escalation study, SA55 will be evaluated for safety, tolerability, and pharmacokinetics. The study is intended to enable future studies of SA55-injection's efficacy in preventing and treating COVID-19.

DETAILED DESCRIPTION:
This is a Phase I, first time in human, randomised, double-blind, placebo-controlled, and dose escalation study.

A Screening Period of up to 14 days (Day -14 through Day 0); A Treatment Period during which participants will be resident at the hospital from Day 0, 1 day before IMP administration (on Day 1) . A Follow up Period lasting 183 days after the IMP dose.

The study will be conducted at a single study centre in Beijing, China.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female 18-65 on the day of enrollment;
* Overall good health condition, with no significant abnormalities during screening and/or pre medication physical examinations;
* Male subjects weighing ≥ 50.0kg; Female subjects with a weight of ≥ 45.0kg and a BMI between 18.0-28.0kg/m2 (including boundary values);
* The subjects and their sexual partners did not have any family planning during the study period, voluntarily took effective contraceptive measures, and did not have plans to donate sperm or eggs; Or for surgical sterilization (female: bilateral fallopian tube ligation, bilateral ovariectomy or hysterectomy; male: vas deferens ligation or vas deferens blockage surgery);
* Volunteer to participate in the experiment, cooperate with the visit, and sign an informed consent form before the start of the study.

Exclusion Criteria:

* Individuals who are known to be allergic to the investigational drug, any component in the preparation, or other similar drugs;
* The test results of hepatitis B B surface antigen (HBsAg), hepatitis C antibody (HCV Ab), HIV antibody (HIV Ab) or Treponema pallidum antibody were positive;
* Suffering from severe neurological disorders (epilepsy, seizures or convulsions) or mental illness, with a family history of mental illness, and neurological and psychiatric problems associated with various organic disorders;
* Abnormal coagulation function (such as coagulation factor deficiency, coagulation disorders, platelet abnormalities) or obvious bruising or coagulation disorders diagnosed by a doctor;
* Other uncontrolled chronic or severe disease history, including but not limited to cardiovascular disease, hematological system disease, liver and kidney disease, digestive system disease, respiratory system disease, malignant tumor, history of major organ transplantation, or any other disease or physiological condition that the researcher believes can interfere with the test results;
* The target injection site (deltoid muscle of the upper arm) may interfere with drug administration or local reaction observation due to skin damage, inflammation, ulcers, rashes, and scars;
* (Female subjects) who are pregnant (including those who have tested positive for pregnancy) or are breastfeeding;
* Have received any SARS-CoV-2 neutralizing antibody injection that is already on the market or in research before screening;
* Participated in clinical trials of other drugs or medical devices within 3 months prior to screening;
* Individuals with a body temperature greater than 37.0 ℃ on the day of medication (Day 1);
* 4 weeks prior to screening for clinically significant acute or chronic disease exacerbations, or a history of surgery;
* It is known that there is a history of SARS CoV-2 infection within 3 months (including positive detection of COVID-19 nucleic acid/antigen during enrollment and screening) or COVID-19 vaccine has been vaccinated;
* Blood donation>400 mL or significant blood loss>400 mL within 3 months prior to medication; Donate plasma or platelets within one month before medication;
* Within the first 6 months of screening, use of immunoglobulins or blood products, immune modulators such as corticosteroids and thymosin α Or blood stimulating drugs;
* Received attenuated live vaccine within 14 days prior to screening, or received subunit or inactivated vaccine within 7 days;
* Those who have used any prescription drugs, over-the-counter drugs, Chinese herbal medicines, and functional vitamins within the first 14 days of screening;
* Smokers who smoke ≥ 5 cigarettes per day within the first 3 months of screening, or who cannot guarantee giving up smoking during the trial period;
* The weekly alcohol consumption in the three months before screening was more than 14 drinking units (1 drinking unit=14g 100% alcohol=360mL beer, or 150mL wine; or 45mL distilled wine/Baijiu), or alcohol abstinence was not allowed during the test, or alcohol breath test was positive before enrollment;
* Have a history of drug abuse or dependence or recreational drug use within 2 years prior to screening, or have a positive urine drug abuse screening before enrollment;
* According to the judgment of the researchers, the subjects have any other factors that are not suitable for participating in clinical trials.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-06-15 (Actual); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of participants with adverse events (AEs) and serious AEs in healthy individuals | 6 months
  The incidence of adverse events (including clinical symptoms and vital signs abnormalities, laboratory examination abnormalities, 12 lead electrocardiogram abnormalities, etc.) and serious adverse events;

SECONDARY OUTCOMES:
Time to reach maximum concentration (Tmax) | 6 months
  Tmax will be assessed after administration of SA55 (IM injection) using noncompartmental methods.
Observed maximum concentration (Cmax) | 6 months
  Cmax will be assessed after administration of SA55 (IM injection) using noncompartmental methods.
Elimination half life (t½) | 6 months
  t½ will be assessed after administration of SA55 (IM injection) using noncompartmental methods.
Systemic clearance (CL) | 6 months
  CL will be assessed after administration of SA55 (IM injection) using noncompartmental methods.
Volume of distribution (Vd) | 6 months
  Vd will be assessed after administration of SA55 (IM injection) using noncompartmental methods.
AUCinf | 6 moths
  AUCinf will be assessed after administration of SA55 (IM injection) using noncompartmental methods.
Anti drug antibody levels (ADA) | 6 months
  To evaluate the serum neutralizing activity of SA55 injection at different time points after administration in healthy individuals. It means anti drug antibody levels (ADA) in serum at different time points

CONTACTS AND LOCATIONS:
Overall Officials: Ronghua Jin, Principal Investigator — Beijing Ditan Hospital
Locations (1):
- Beijing Ditan Hospital Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhou Y, Meng X, Li J, Zeng G, Wang J, Cao Y, Hu C, Jin R. Safety, tolerability, and pharmacokinetics of anti-SARS-CoV-2 monoclonal antibody SA55 injection in healthy participants. Antimicrob Agents Chemother. 2025 Aug 6;69(8):e0056825. doi: 10.1128/aac.00568-25. Epub 2025 Jul 17. PMID 40673766